CLINICAL TRIAL: NCT00149513
Title: King County Lung Injury Project: Survivor Outcome Study (KCLIP:SOS)
Brief Title: Post-Hospital Case Management to Improve Clinical Outcomes in Individuals Requiring Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Parsons, Assistant Professor, SOM: Department of Medicine: Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25934; P50HL073996 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Targeted nurse case management
  Interventions: Behavioral: Targeted Case Management
- 2 (Active Comparator): Usual Care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Targeted Case Management — A nurse case manager will assess and follow intervention arm subjects for six months. Nurse case manager will help subjects acquire needed community health services.
  Arms: 1
Behavioral: Usual care — Participants will receive usual care.
  Arms: 2

SUMMARY:
King County Lung Injury Project: Survivor Outcome Study (KCLIP:SOS) is a randomized trial for individuals who have survived prolonged mechanical ventilation (5 days or more). The objective is to enroll individuals who are likely to have impaired health status resulting from prolonged critical illness but whose long term prognosis is good. Such individuals are most likely to benefit from the study intervention of case management targeted at post intensive care complications.

KCLIP:SOS will test whether an outpatient intervention based on a nurse using a targeted case management tool can reduce patient morbidity and improve quality of life in the 6 months following hospital discharge. This intervention will be compared to usual post-hospital care.

DETAILED DESCRIPTION:
BACKGROUND:

The purpose of this study is to understand individuals' physical and emotional conditions and concerns after being ventilated in the hospital. Modern hospital care helps many people survive even if they are on ventilators for long periods of time. Some individuals who leave the hospital after this kind of intensive care suffer from depression, post-traumatic stress disorder, muscle weakness, tiredness or breathing difficulties that may decrease their quality of life. Doctors know little about finding and treating these problems in survivors of mechanical ventilation.

DESIGN NARRATIVE:

Participants will be randomly assigned in blocks of 10 (5 participants to usual care and 5 participants to case management) for home or skilled nursing facility discharges. The Outcome Assessors (the interviewers collecting outcomes data) will be blinded to group assignment.

Primary outcome: All participants will have a baseline interview soon after hospital discharge and a final interview at the end of the 6-month intervention period (outcome assessments). All subjects will be asked to keep a diary/journal of their medical appointments, health services, and medications. Participants will be called once a month to collect this information.

Key secondary outcomes: Case management participants will be contacted by the nurse case manager who will provide follow-up care for 6 months. At the end of the study, interview results will be sent to the personal physician of the usual care participants so that appropriate care can follow.

ELIGIBILITY:
Inclusion Criteria:

* On a ventilator for 5 or more days
* Expected to survive the 6 months post-hospital discharge period
* Lives in the SOS zip code area (King, Pierce and Snohomish counties)

Exclusion Criteria:

* Severe pre-hospital health conditions
* Lack of availability for follow-up (e.g. homeless, chronic substance abuse)
* Non-English speakers
* Severe psychiatric issues
* Need for special rehabilitation services not available in the intervention
* Predicted survival of less than 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Scores for quality of life measures | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Rubenfeld, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States